CLINICAL TRIAL: NCT03942211
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study in Participants With Sarcoidosis-Associated Pulmonary Hypertension (SAPH) to Assess the Efficacy and Safety of Oral Selexipag.
Brief Title: A Study in Participants With Sarcoidosis-associated Pulmonary Hypertension (SAPH) to Assess the Efficacy and Safety of Oral Selexipag
Acronym: SPHINX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to prematurely terminate the study due to the lower-than-expected recruitment rate
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-065D301; 2018-004887-74 (EudraCT Number)
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Sarcoidosis-associated Pulmonary Hypertension
Keywords: selexipag, sarcoidosis, pulmonary hypertension
MeSH Terms: conditions — Sarcoidosis; Hypertension, Pulmonary | interventions — selexipag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selexipag 200 micro gram (μg) (Experimental): Study intervention will be up-titrated to allow each participant to reach their individual maximum tolerated dose (iMTD), in the range of 200 μg to1600 μg (ie, 1 to 8 tablets) twice daily/once daily. Dosing frequency will be twice daily, except for participants with moderate hepatic impairment (Child-Pugh Class B) or who are concomitantly taking (a) moderate CYP2C8 inhibitor(s), who receive study intervention once daily. The dose will be up-titrated by the investigator/delegate in 200 μg twice daily/once daily increments at weekly intervals during scheduled TCs until reaching the iMTD. If the dose regimen is not well tolerated or symptoms cannot be fully managed with symptomatic treatment, the duration of the titration step can be prolonged to 2 weeks. If needed, the dose can be reduced by 200 μg twice daily/once daily.
  Interventions: Drug: Selexipag
- Placebo (Placebo Comparator): The comparator will be administered similarly to the experimental intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selexipag — Oral tablets containing 200 µg of selexipag. Depending on the iMTD, participants will receive 1 (200 µg) to 8 (1600 µg) tablets at each administration
  Other Names: JNJ-678896049; ACT-293987
  Arms: Selexipag 200 micro gram (μg)
Drug: Placebo — Oral tablets without active compound. Participants can receive 1 to 8 tablets at each administration.
  Arms: Placebo

SUMMARY:
Oral selexipag is commercially available in several countries for the treatment of a particular group of pulmonary hypertension (PH) called pulmonary arterial hypertension (PAH). The aim of the present study is to investigate whether selexipag could be helpful to treat patients with another form of PH called sarcoidosis-associated pulmonary hypertension (SAPH).

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a pathophysiological disorder that may involve multiple clinical conditions and can complicate several cardiovascular and respiratory diseases. Sarcoidosis is a multisystemic disorder that is characterized by non-caseating granulomas which are present in multiple tissues, particularly in the lung and lymphatic system. Severe untreated pulmonary hypertension (PH) carries a poor prognosis and is associated with higher mortality in participants with interstitial lung diseases and sarcoidosis. While there is no approved treatment for SAPH, PH-specific treatments are frequently used. Selexipag is a selective, orally available and long-acting non-prostanoid agonist of the prostacyclin receptor (prostacyclin [IP] receptor) for the treatment of patients with PAH. The rationale for this study is based on the unmet medical need for new therapeutic options for patients with SAPH and is supported by the established efficacy and safety of selexipag in the PAH indication, the shared pathomechanism between SAPH and PAH, and the available data on the efficacy and safety of PH-specific therapies in SAPH. This study consists of screening period, main observation period and double blind extension period and safety follow-up period. The duration of individual participation in the study will be different for each individual participant (between approximately 15 months and up to approximately 3.5 years) and will depend on the time of each participant's individual date of entering the study and the total recruitment time. The efficacy assessments include right heart catheterization (RHC), assessment of exercise capacity, dyspnea, pulmonary function tests, etc. Safety and tolerability will be evaluated throughout the study and includes review of concomitant medications and adverse events (AEs), clinical laboratory tests, 12-lead electrocardiogram (ECG), vital signs, physical examination, and pregnancy testing.

ELIGIBILITY:
Main Inclusion Criteria:

* Confirmed diagnosis of sarcoidosis as per American Thoracic Society (ATS) criteria
* Sarcoidosis-associated precapillary PH, confirmed by RHC (at rest) within 90 days prior to randomization.
* PH severity according to modified WHO FC II-IV at Screening and randomization; participants in WHO FC IV must be in a stable condition and able to perform a 6MWT.
* Either not receiving treatment with PH-specific treatment or oral PH-specific monotherapy (ie, riociguat or PDE5i or ERA); if on oral PH-specific monotherapy then treatment had to be stable (ie, no introduction of new therapies or changes in dose) for at least 90 days prior to both and the RHC qualifying for enrollment and randomization
* Stable sarcoidosis treatment regimen, ie, no new specific anti-inflammatory treatment for sarcoidosis for at least 90 days, and stable dose(s) for at least 30 days prior to both the RHC qualifying for enrollment and randomization
* 6-minute walk distance (6MWD) greater than or equal to (>=) 50 meters both at Screening and at the time of randomization. Participants can use their usual walking aids during the test (example, cane, crutches). The same walking aid should be used for all 6-minute walk test (6MWTs). Walkers are not allowed
* Forced Vital Capacity (FVC) greater than (>) 50 percent (%) and Forced Expiratory Volume (in 1 second) (FEV1) > 50% of predicted at Screening
* Diffusing capacity of the lung for carbon monoxide (DLCO) >= 40% of predicted. If DLCO less than (<) 40% of predicted, the extent of emphysema should not be greater than that of fibrosis as assessed by high resolution computerized tomography (CT) scan
* Women of childbearing potential must have a negative pregnancy test at screening and randomization, must agree to undertake monthly urine pregnancy tests, and to practice an acceptable method of contraception and agreeing to remain on an acceptable method while receiving study intervention and until 30 days after last dose of study intervention
* A woman only using hormonal contraceptives must have been using this method for at least 30 days prior to randomization

Main Exclusion Criteria:

* PH due to left heart disease (PAWP >15 mmHg).
* History of left heart failure (LHF) as assessed by the investigator including cardiomyopathies, and cardiac sarcoidosis, with a left ventricular ejection fraction (LVEF) <40%.
* Treatment with prostacyclin, prostacyclin analogues or IP receptor agonists (ie, selexipag) within 90 days prior to randomization and/or prior to the RHC qualifying for enrollment, except those given at vasodilator testing during RHC.
* SBP <90 mmHg at Screening or at randomization.
* Included on a lung transplant list or planned to be included until Visit 6 / Week 39.
* Change in dose or initiation of new diuretics and/or calcium channel blockers within 1 week prior to RHC qualifying for enrollment.
* Any condition for which, in the opinion of the investigator, participation would not be in the best interests of the participant (eg, compromise well-being), or that could prevent, limit, or confound the protocol-specified assessments.
* Any acute or chronic impairment that may influence the ability to comply with study requirements such as to perform RHC, a reliable and reproducible 6MWT, or lung function tests.
* Any other criteria as per selexipag Summary of Product Characteristics (SmPC)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Zimmermann, Study Director — Actelion
Locations (38):
- United States (8):
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - LSU Health Sciences Center New Orleans, New Orleans, Louisiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina (MUSC) - College of Medicine (COM), Charleston, South Carolina
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Brazil (3):
  - Secretaria da Saude do Estado do Ceara - Hospital Doutor Carlos Alberto Studart Gomes, Fortaleza
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (5):
  - Hôpital Avicenne, Bobigny
  - GH est - Hôpital Cardiovasculaire et Pneumologie Louis Pradel, Bron
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hopital Nord, Marseille
  - CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Thoraxklinik Heidelberg, Heidelberg
  - Universitatsklinikum Schleswig Holstein, Lübeck
  - Universitaetsklinikum Regensburg, Regensburg
  - RBK Lungenzentrum Stuttgart am Robert-Bosch-Krankenhaus, Stuttgart
  - Klinikum Würzburg Mitte gGmbH Standort Missioklinik, Würzburg
- Italy (5):
  - Ospedale S.Giuseppe, Gruppo MultiMedica, Milan
  - Fondazione Maugeri Montescano, Pavia
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - Universita Cattolica del Sacro Cuore - Fondazione Policlinico Universitario 'A. Gemelli', Roma
  - A.O.U. Città della Salute e della Scienza, Torino
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - Sint Antonius Ziekenhuis, Nieuwegein
- Spain (2):
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. Univ. Marques de Valdecilla, Santander
- United Kingdom (2):
  - Royal Free Hospital, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Actelion is a Janssen pharmaceutical company of Johnson & Johnson. The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Selexipag 200 Micrograms (mcg): Participants received a single oral tablet of selexipag 200 mcg on Day 1. The dose was up-titrated by the investigator/delegate at weekly intervals to allow each participant to reach their individual maximum tolerated dose (iMTD), in the range of 200 mcg to 1600 mcg (that is, 1 to 8 tablets) twice daily from Day 2 to Week 12 or until reaching iMTD. From Week 12 onwards, participants received their iMTD of selexipag orally twice daily till end of treatment (up to 456 days). For participants with moderate hepatic impairment (Child-Pugh Class B) or who were concomitantly taking moderate CYP2C8 inhibitor(s) the dosing frequency was once daily.
- Placebo: Participants received placebo matching to selexipag 1 to 8 tablets twice daily from Day 1 till end of treatment (up to 456 days). For participants with moderate hepatic impairment (Child-Pugh Class B) or who were concomitantly taking moderate CYP2C8 inhibitor(s) the dosing frequency was once daily.
Period: Overall Study
Arm/Group | Selexipag 200 Micrograms (mcg) | Placebo
Started | 6 | 4
Completed | 0 | 0
Not Completed | 6 | 4
Not completed — Death | 1 | 0
Not completed — Study terminated by sponsor | 5 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selexipag 200 Micrograms (mcg) | Placebo | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (14.53) | 68.5 (2.38) | 60.4 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  France | 0 | 1 | 1
  Germany | 4 | 0 | 4
  Spain | 1 | 1 | 2
  United Kingdom | 1 | 0 | 1
  United States | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Vascular Resistance (PVR) up to Week 26
Description: PVR represents the resistance against which the right ventricle needs to pump. PVR was determined by right heart catheterization (RHC). It was measured as the ratio of the PVR value post-treatment initiation up to Week 26 (post) versus the PVR value pre-treatment initiation at baseline (pre), expressed as a percentage of baseline value. The baseline reference value for PVR was based on the last RHC performed prior to study intervention initiation. PVR was calculated as 80*(mean pulmonary arterial pressure - pulmonary artery wedge pressure) divided by cardiac output. As specified in the statistical analysis plan, data was not planned to be summarized for this outcome measure and only individual participant wise data was collected.
Time Frame: Baseline up to Week 26
Population: Randomized analysis set included all participants assigned to the study intervention. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants randomized and analyzed in respective treatment arm. Here, 'n' (number analyzed)=0 signifies that the participant was not randomized in that treatment arm.
Measure: Number; unit: percentage of baseline PVR
Arm/Group | Selexipag 200 Micrograms (mcg) | Placebo
Number analyzed (Participants) | 5 | 3
percentage of baseline PVR
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 89.0
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 201
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 56
  Participant 4: number analyzed (Participants) | 1 | 0
  Participant 4 | 88 |
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 100 |
  Participant 6: number analyzed (Participants) | 1 | 0
  Participant 6 | 47.0 |
  Participant 7: number analyzed (Participants) | 1 | 0
  Participant 7 | 82.0 |
  Participant 8: number analyzed (Participants) | 1 | 0
  Participant 8 | 86.0 |

ADVERSE EVENTS:
Time Frame: From Day 1 up to 456 days
Description: Safety assessments were based on the safety analysis set which included all participants who received at least one dose of study intervention.
Arm/Group | Selexipag 200 Micrograms (mcg) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/4
Other Adverse Events (participants affected / at risk) | 6/6 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag 200 Micrograms (mcg) (N=6) | Placebo (N=4)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag 200 Micrograms (mcg) (N=6) | Placebo (N=4)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (13) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sputum Purulent (Infections and infestations) | 0 (0) | 1 (1)
Injection Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0)
Glycosylated Haemoglobin Increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0)
Mean Cell Haemoglobin Increased (Investigations) | 1 (1) | 0 (0)
Mean Cell Volume Increased (Investigations) | 1 (1) | 0 (0)
N-Terminal Prohormone Brain Natriuretic Peptide Increased (Investigations) | 1 (1) | 0 (0)
Neutrophil Count Increased (Investigations) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Red Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (2) | 0 (0)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 5 (11) | 1 (2)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Papulopustular Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cyanosis (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
All planned efficacy analyses could not be performed due to early termination of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03942211/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03942211/SAP_001.pdf